CLINICAL TRIAL: NCT04625049
Title: Does Microglial Activation Promote Lesion Growth and Progression Among Multiple Sclerosis Patients
Acronym: FUP-MS
Status: Enrolling by invitation | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FUP-MS
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The purpose of this study is to assess whether increased microglial activation (measured using TSPO-PET) at lesion rim is associated with more rapid lesion growth during 10 year follow up.

DETAILED DESCRIPTION:
Objective: To evaluate individual MS lesions and their growth during a total of 10 year follow-up after initial positron emission tomography (PET) -imaging with PK11195 or TMSX radioligands.

Background: Focal inflammatory lesions in the white and grey matter of the central nervous system represent the best characterized pathological phenomena of MS disease. Some MS lesions slowly expand over time. Neuropathological studies have detected inflammatory rim formed by activated microglia cells around some MS lesions and it has been suggested that the presence of the inflammatory rim could predict lesion expansion. Our hypothesis is that the lesions with higher TSPO or TMSX radioligand binding at the initial PET scan will expand more during the total of 10-year follow up compared to those lesions with lower radioligand binding. This longitudinal follow-up study will provide a more complete picture of the association of the innate immune cell activation, lesion growth and disease progression.

Study population: The research will recruit approximately 100 MS-patients who have taken part to our previous PET-imaging MS studies in Turku PET centre. The research interventions will consist of magnetic resonance imaging (MRI) scans, blood sampling, clinical neurological evaluation and patient-reported outcome measures (filling forms).

ELIGIBILITY:
Inclusion Criteria:

* Participation to a previous PET imaging study of Airas group
* MS diagnosis

Exclusion Criteria:

* Patients with other neurodegenerative disease than MS
* Contraindication to MR scan investigations
* Patients with claustrophobia, or a history of moderate to severe anxiety disorder or panic attacks (which could potentially lead to preterm termination of the imaging)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research will recruit MS-patients who have taken part to our previous PET-imaging MS studies in Turku PET centre. The research interventions will consist of MRI scans, blood sampling, clinical neurological evaluation and patient-reported outcome measures (filling forms).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Correlation of the lesion volume changes to the microglial activity at the initial positron emission tomography imaging | Baseline (initial PET), 3, 5, 7 and 10 years
  Correlation of the lesion volume changes in the magnetic resonance imaging to the microglial activity at the initial PET imaging

SECONDARY OUTCOMES:
magnetic resonance imaging metrics | Baseline (initial PET), 3, 5, 7 and 10 years
  To evaluate whole brain, white matter, gray matter volumes during follow-up
Multiple Sclerosis Composite Score | Baseline (initial positron emission tomography), 3, 5, 7 and 10 years
  Multiple Sclerosis Composite Score which consists of three assessments of walking speed, processing speed and finger dexterity. The scores are combined to provide a Z-score. Lower scores represent greater abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, Principal Investigator — Turku University Hospital, Division of Clinical Neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland